CLINICAL TRIAL: NCT03954106
Title: Prospective, Multicenter, Open-Label, Single Arm, Phase 2 Study to Evaluate the Safety and Efficacy of Defibrotide in the Prevention of Chimeric Antigen Receptor-T-cell-associated Neurotoxicity in Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma Receiving Axicabtagene Ciloleucel (Yescarta®)
Brief Title: A Safety and Efficacy Study of Defibrotide in the Prevention of Chimeric Antigen Receptor-T-cell-associated Neurotoxicity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary endpoint would unlikely to be met based on the unplanned interim assessment on the first 20 efficacy evaluable patients.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JZP395-201
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: DLBCL; Neurotoxicity Syndromes
Keywords: CAR-T
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — defibrotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Defibrotide (Experimental): Part 1 (lead-in phase) will evaluate a 2.5 mg/kg/dose regimen before escalating to a 6.25 mg/kg/dose regimen.
  After the Safety Assessment Committee establishes the recommended phase 2 dose based on dose-limiting toxicities during Part 1, Part 2 will enroll subjects at the recommended phase 2 dose.
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — * Part 1: Defibrotide 2.5 mg/kg/dose or 6.25 mg/kg/dose once daily as a single dose on CAR-T Day -5, -4, and -3 before lymphodepletion, then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7).
  * Part 2 Recommended Phase 2 Dose: Defibrotide 6.25 mg/kg/dose once daily as a single dose on CAR-T Day -5, -4, and -3 before lymphodepletion, then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7).

SUMMARY:
This is a prospective, open-label, single-arm study evaluating the safety and efficacy of defibrotide for the prevention of CAR-T-associated neurotoxicity in subjects with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) receiving Yescarta.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age at signing of informed consent.
2. Subject must be diagnosed with relapsed or refractory DLBCL (including DLBCL not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma) and scheduled to receive treatment with Yescarta.
3. Female subjects of childbearing potential who are sexually active and male subjects who are sexually active and have female partners of childbearing potential must agree to use a highly effective method of contraception with their partners during exposure to defibrotide and for 30 days after the last dose of defibrotide.
4. Subject must be able to understand and sign written informed consent.

Exclusion Criteria:

1. Subject is currently receiving dialysis or expected to receive dialysis.
2. Subject has used any investigational anticancer agent within 3 weeks prior to the first dose of defibrotide, or is using or plans to use any investigational agent during the study.
3. Subject has previously been treated with CAR-T therapy.
4. Hemodynamic instability requiring vasopressors or uncontrolled hypertension with persistent systolic blood pressure > 180.
5. Subject has clinically significant active bleeding, history of intracranial bleeding, or is at risk for intracranial bleeding as determined by the Investigator.
6. Subject plans to use any medication that increases the risk of bleeding.
7. Subject is pregnant or lactating and does not agree to stop breastfeeding.
8. Subject has a known history of hypersensitivity to defibrotide or any of the excipients.
9. Subject has primary CNS lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mayo Clinic, Phoenix, Arizona
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Jacobson CA, Rosenthal AC, Arnason J, Agarwal S, Zhang P, Wu W, Amber V, Yared JA. A phase 2 trial of defibrotide for the prevention of chimeric antigen receptor T-cell-associated neurotoxicity syndrome. Blood Adv. 2023 Nov 14;7(21):6790-6799. doi: 10.1182/bloodadvances.2023009961. PMID 37399456
- [Derived] Danish H, Santomasso BD. Neurotoxicity Biology and Management. Cancer J. 2021 Mar-Apr 01;27(2):126-133. doi: 10.1097/PPO.0000000000000507. PMID 33750072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient disposition was assessed in the Safety Analysis Set (N=25) which was comprised of the Part 1: Defibrotide 2.5 mg/kg/dose (n=4) and the combined Part 1: Defibrotide 6.25 mg/kg/dose and Phase 2: RP2D 6.25 mg/kg/dose (n=21). The patient disposition is reported in this format as per the Statistical Analysis Plan.
Groups:
- Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose: Participants who received the safety (lead in) dose of 2.5 mg/kg/dose defibrotide once daily as a single dose on CAR-T Day -5, -4, and -3 prior to lymphodepletion and then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7).
- Phase 2: RP2D, Defibrotide 6.25 mg/kg/Dose: Participants who received the recommended phase 2 dose of 6.25 mg/kg/dose defibrotide once daily as a single dose on CAR-T Day -5, -4, and -3 prior to lymphodepletion and then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7).
Period: Part 1: Safety Lead In Phase
Arm/Group | Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose | Phase 2: RP2D, Defibrotide 6.25 mg/kg/Dose
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0
Period: Phase 2: Treatment at RP2D
Arm/Group | Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose | Phase 2: RP2D, Defibrotide 6.25 mg/kg/Dose
Started | 0 | 21
Completed | 0 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographics were assessed in the Safety Analysis Set (N=25) which was comprised of the Part 1: Defibrotide 2.5 mg/kg (n=4) and the combined Part 1: Defibrotide 6.25 mg/kg and Phase 2: RP2D 6.25 mg/kg (n=21). The baseline demographics are reported in this format as per the Statistical Analysis Plan.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose | Phase 2: RP2D, Defibrotide 6.25 mg/kg/Dose | Total
Number analyzed (Participants) | 4 | 21 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 7 | 9
  >=65 years | 2 | 14 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 3 | 14 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 21 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 21 | 25

OUTCOME MEASURES:

1. Primary Outcome: Incidence of CAR-T-associated Neurotoxicity of Any Grade, Defined by CTCAE v5.0 by CAR-T Day +30
Description: The primary efficacy endpoint was the incidence of CAR-T-associated neurotoxicity of any grade defined by CTCAE v5.0 by CAR-T Day +30. The results report the estimated percentage of participants with no CAR-T-associated neurotoxicity of any grade, defined by CTCAE v5.0, which incorporated the 2 stage design.
Time Frame: By CAR-T Day +30
Population: The Efficacy Evaluable Analysis Set consisted of all participants in the Enrolled (RP2D) Analysis Set who received at least 18 doses (of all 35) of defibrotide and either developed CAR-T-associated neurotoxicity on or before CAR-T Day +30; OR completed the CAR-T Day +30 neurological assessment and discontinued defibrotide due to CAR-T-associated neurotoxicity before receiving 18 doses of defibrotide.
  Yescarta infusion must NOT have been delayed by more than 2 days from the original schedule.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Stage 1: Defibrotide, 6.25 mg/kg/Dose: Participants who either received the safety (lead in) dose of 6.25 mg/kg/dose defibrotide in Part 1 (n=4) or received the RP2D of 6.25 mg/kg/dose defibrotide in Part 2 (n=6) once daily as a single dose on CAR-T Day -5, -4, and -3 prior to lymphodepletion and then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7). Stage 1 participants are the first 10 efficacy evaluable participants.
- Stage 2: Defibrotide, 6.25 mg/kg/Dose: Participants who received the RP2D of 6.25 mg/kg/dose defibrotide in Part 2 (n=10) once daily as a single dose on CAR-T Day -5, -4, and -3 prior to lymphodepletion and then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7). Stage 2 participants include the additional efficacy evaluable participants enrolled after the completion of Stage 1.
- Overall: Defibrotide, 6.25 mg/kg/Dose: All participants who received 6.25 mg/kg/dose defibrotide once daily as a single dose on CAR-T Day -5, -4, and -3 prior to lymphodepletion and then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7) in Stage 1 and Stage 2.
Arm/Group | Stage 1: Defibrotide, 6.25 mg/kg/Dose | Stage 2: Defibrotide, 6.25 mg/kg/Dose | Overall: Defibrotide, 6.25 mg/kg/Dose
Number analyzed (Participants) | 10 | 10 | 20
percentage of participants | 50 [NA to NA] — As per the Statistical Analysis Plan, confidence intervals (CIs) were not calculated for the primary outcome for Stage 1 or Stage 2. CIs were only calculated for the Overall: Defibrotide 6.25 mg/kg/dose group. | 50 [NA to NA] — As per the Statistical Analysis Plan, confidence intervals (CIs) were not calculated for the primary outcome for Stage 1 or Stage 2. CIs were only calculated for the Overall: Defibrotide 6.25 mg/kg/dose group. | 51 [36 to 66]

2. Secondary Outcome: Incidence of CAR-T-Associated Neurotoxicity Grade 3 or Greater Defined by CTCAE v5.0 by CAR-T Day +30
Description: The secondary efficacy endpoint was the incidence of CAR-T-associated neurotoxicity Grade 3 or greater defined by CTCAE v5.0 by CAR-T Day +30. The results report the estimated percentage of participants with no CAR-T-associated neurotoxicity (Grade 3 or greater defined by CTCAE v5.0) by CAR-T Day +30.
Time Frame: By CAR-T Day +30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Defibrotide, 6.25 mg/kg/Dose | Stage 2: Defibrotide, 6.25 mg/kg/Dose | Overall: Defibrotide, 6.25 mg/kg/Dose
Number analyzed (Participants) | 10 | 10 | 20
percentage of participants | 80 | 70 | 75

3. Secondary Outcome: Incidence of CAR-T-Associated Neurotoxicity of Any Grade According to the ASBMT Consensus Grading System by CAR-T Day +30
Description: The secondary efficacy endpoint was the incidence of CAR-T-associated neurotoxicity of any grade according to ASBMT consensus grading system by CAR-T Day +30. The results report the estimated percentage of participants with no CAR-T-associated neurotoxicity by CAR-T Day +30 summarized descriptively by any grade according to the ASBMT consensus grading system.
Time Frame: By CAR-T Day +30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Defibrotide, 6.25 mg/kg/Dose | Stage 2: Defibrotide, 6.25 mg/kg/Dose | Overall: Defibrotide, 6.25 mg/kg/Dose
Number analyzed (Participants) | 10 | 10 | 20
percentage of participants | 0 | 0 | 0

4. Secondary Outcome: Incidence of CAR-T-Associated Neurotoxicity of Grade 3 or Greater According to the ASBMT Consensus Grading System by CAR-T Day +30
Description: The secondary efficacy endpoint was the incidence of CAR-T-associated neurotoxicity grade 3 or greater according to ASBMT consensus grading system by CAR-T Day +30. The results report the estimated percentage of participants with no CAR-T-associated neurotoxicity by CAR-T Day +30 summarized descriptively by grade 3 or greater according to the ASBMT consensus grading system.
Time Frame: By CAR-T Day +30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Defibrotide, 6.25 mg/kg/Dose | Stage 2: Defibrotide, 6.25 mg/kg/Dose | Overall: Defibrotide, 6.25 mg/kg/Dose
Number analyzed (Participants) | 10 | 10 | 20
percentage of participants | 90 | 70 | 80

5. Secondary Outcome: Incidence of Cytokine Release Syndrome (CRS) of Any Grade According to the ASBMT Consensus Grading System by CAR-T Day +30
Description: The secondary efficacy endpoint was the incidence of cytokine release syndrome (CRS) of any grade according to ASBMT consensus grading system by CAR-T Day +30. The results report the estimated percentage of participants with no CRS any grade according to ASBMT criteria and was summarized descriptively using the ASBMT consensus grading system by CAR-T Day +30.
Time Frame: By CAR-T Day +30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1: Defibrotide, 6.25 mg/kg/Dose | Stage 2: Defibrotide, 6.25 mg/kg/Dose | Overall: Defibrotide, 6.25 mg/kg/Dose
Number analyzed (Participants) | 10 | 10 | 20
percentage of participants | 10 | 20 | 15

6. Secondary Outcome: Use of High Dose Steroid By CAR-T Day +30
Description: The percentage of participants using high dose steroids was summarized descriptively. The use of high dose steroids was defined as a dose of dexamethasone of at least 7.5 mg/day or equivalent. Only the Overall Defibrotide: 6.25 mg/kg/dose group was analyzed for this outcome.
Time Frame: By CAR-T Day +30
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Overall: Defibrotide, 6.25 mg/kg/Dose
Number analyzed (Participants) | 20
percentage of participants | 45

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were recorded from the time the subject signed informed consent until the final study visit or Early Termination (ET).
Description: Adverse events (AEs), SAEs, and all-cause mortality were assessed in the Safety Analysis Set (N=25) which comprised of the Part 1: Defibrotide 2.5 mg/kg/dose (n=4) and the combined Part 1: Defibrotide 6.25 mg/kg/dose and Phase 2: RP2D 6.25 mg/kg/dose (n=21). The safety data are reported in this format as per the Statistical Analysis Plan.
Groups:
- Phase 2: RP2D, 6.25 mg/kg/Dose: Participants who received the recommended phase 2 dose of 6.25 mg/kg/dose defibrotide once daily as a single dose on CAR-T Day -5, -4, and -3 prior to lymphodepletion and then every 6 hours daily for 8 days (CAR-T Day 0 to Day 7).
Arm/Group | Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose | Phase 2: RP2D, 6.25 mg/kg/Dose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/21
Serious Adverse Events (participants affected / at risk) | 4/4 | 9/21
Other Adverse Events (participants affected / at risk) | 4/4 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose (N=4) | Phase 2: RP2D, 6.25 mg/kg/Dose (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Safety Lead-In, Defibrotide 2.5 mg/kg/Dose (N=4) | Phase 2: RP2D, 6.25 mg/kg/Dose (N=21)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 6 (9)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 10 (25)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (8)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (3)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 6 (6)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 4 (6)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 11 (16)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 12 (14)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 14 (14)
Vommiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 10 (13)
Fatigue (General disorders) | 1 (1) | 12 (13)
Gait disturbance (General disorders) | 0 (0) | 4 (4)
Generalized oedema (General disorders) | 1 (1) | 0 (0)
Localized oedema (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 5 (6)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (7) | 17 (48)
Cytokine release syndrome (Immune system disorders) | 3 (4) | 15 (27)
Candida infection (Infections and infestations) | 0 (0) | 3 (4)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 3 (3)
Blood sodium decrreased (Investigations) | 0 (0) | 2 (2)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1)
Blood urea decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2)
Clostridium test (Investigations) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (5) | 1 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 7 (8)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (4) | 6 (11)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 5 (6)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Muscle Spasma (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6)
Aphasia (Nervous system disorders) | 1 (1) | 4 (6)
Atazia (Nervous system disorders) | 0 (0) | 1 (1)
Cognative disorder (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 6 (8)
Dysarthria (Nervous system disorders) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 2 (2) | 10 (15)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Neurotoxicity (Nervous system disorders) | 0 (0) | 7 (16)
Presyncope (Nervous system disorders) | 1 (1) | 2 (4)
Tremor (Nervous system disorders) | 1 (2) | 11 (17)
Agitation (Psychiatric disorders) | 1 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 2 (3) | 7 (24)
Delirium (Psychiatric disorders) | 0 (0) | 3 (3)
Dysphemia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress unrinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 5 (5)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Penile haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoes (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (10)
Laryngeal haemorrage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tachypnoes (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (6) | 14 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2019-02-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT03954106/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT03954106/SAP_001.pdf